CLINICAL TRIAL: NCT05856552
Title: The Health and Social Consequences of Depression Among the Elderly: Evidence From India
Brief Title: The Health and Social Consequences of Depression Among the Elderly
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Bureau of Economic Research, Inc. (Other)
Collaborators: Abdul Latif Jameel Poverty Action Lab (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 23003
Record Dates: First submitted 2023-04-24; First posted 2023-05-12 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Depression; Functional Impairment
Keywords: Elderly; India; CBT; Group activities; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CBT home visits (Experimental): Community resource persons will visit the elderly women once per week to deliver cognitive behavioral therapy for six weeks, followed by 3 monthly boosters. For half the experimental sample, the boosters will be an ongoing monthly intervention beyond the initial 6-week period.
  Interventions: Behavioral: CBT
- CBT home visits and group activities (Experimental): Community resource persons will visit the elderly women once per week to deliver cognitive behavioral therapy for six weeks, followed by 3 monthly boosters. The elderly women will also be invited to join weekly hour-long group activities for 12 weeks. Group activities will be administered by community resource persons in community spaces. For half of the experimental sample, the group activities will be an ongoing weekly intervention beyond the initial 12-week period, and the CBT booster sessions will be administered monthly after the initial 6-week period.
  Interventions: Behavioral: CBT; Behavioral: Group Activities
- Control (No Intervention): Control group
- Group activities (Experimental): The elderly women will be invited to join weekly hour-long group activities for 12 weeks. Group activities will be administered by community resource persons in community spaces. For half of the experimental sample, the group activities will be an ongoing weekly intervention beyond the initial 12-week period.
  Interventions: Behavioral: Group Activities

INTERVENTIONS:
Behavioral: CBT — Cognitive behavioral therapy delivered by community resource persons via home visits.
  Arms: CBT home visits; CBT home visits and group activities
Behavioral: Group Activities — Weekly hour-long group activities delivered by community resource persons in community spaces.
  Arms: CBT home visits and group activities; Group activities

SUMMARY:
Mental illnesses often go undiagnosed or untreated in low-income settings. Mental health care may be especially important for the elderly - events in the lives of the elderly, like illnesses or deaths of peers, may put these individuals at high risk of mental illness. The study will constitute a randomized controlled trial aimed at reducing depression among elderly women. Through two interventions, the investigators will aim to improve women elder's outlook on life and relationships through cognitive behavioral therapy (CBT) and facilitated group activities. There will be a total of four treatment arms: one for CBT during home visits, one for facilitated group activities, one for both, and a control group receiving neither the CBT nor facilitated group activities. All activities will be delivered by lay government community volunteers. Randomization for group activities will be at the village level, and randomization for CBT will be at the individual-level within each village. Investigators will track outcomes of the elderly at two points in time: immediately after the main 12-week intervention period and 6 months after the main intervention period.

ELIGIBILITY:
Inclusion Criteria:

* At least 55 years of age
* Women

Exclusion Criteria:

* Those with hearing, speech or mental impairment

Min Age: 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5370 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Depression Score | Assessed at 0 months after the intervention
  The geriatric depression scale short form (GDS-15) is used. Participants are asked 15 yes/no questions: if they are satisfied with their lives, have dropped activities and interests, feel their life is empty, often get bored, are in good spirits most of the time, are afraid that something bad is going to happen to them, feel happy most of the time, often feel hopeless, prefer to stay at home, rather than going out and doing new things, have more problems with memory, think it is wonderful to be alive, feel worthless, feel full of energy, feel lonely, feel their situation is hopeless, think that most people are better off than they are. Responses will be summed over these questions (scale of 0-15) with answers coded such as 1 indicates a depressive symptom for that question and 0 otherwise.
Depression Score | Assessed at 6 months after the intervention
  The geriatric depression scale short form (GDS-15) is used. Participants are asked 15 yes/no questions: if they are satisfied with their lives, have dropped activities and interests, feel their life is empty, often get bored, are in good spirits most of the time, are afraid that something bad is going to happen to them, feel happy most of the time, often feel hopeless, prefer to stay at home, rather than going out and doing new things, have more problems with memory, think it is wonderful to be alive, feel worthless, feel full of energy, feel lonely, feel their situation is hopeless, think that most people are better off than they are. Responses will be summed over these questions (scale of 0-15) with answers coded such as 1 indicates a depressive symptom for that question and 0 otherwise.
Difficulty in performing daily activities/Functional impairment score | Assessed at 0 months after the intervention
  The 12-item WHO Disability Assessment Schedule 2.0 questionnaire is used. Participants will be asked the level of difficulty they have in doing each of the following tasks in the past 30 days due to health conditions: standing for long periods such as 30 minutes, walking a long distance (such as 1km), concentrating for 10 minutes, learning a new task like getting to a new place, washing whole body, getting dressed, taking care of household responsibilities, doing day-to-day work, dealing with people they do not know, maintaining a friendship, being emotionally affected by health problems, and joining in community activities. The scale is from 0-4, with 0 being no difficulty, 1 mild, 2 moderate, 3 severe, and 4 cannot do. The scores will be summed to create a cumulative score on a 0-48 scale.
Difficulty in performing daily activities/Functional impairment score | Assessed at 6 months after the intervention
  The 12-item WHO Disability Assessment Schedule 2.0 questionnaire is used. Participants will be asked the level of difficulty they have in doing each of the following tasks in the past 30 days due to health conditions: standing for long periods such as 30 minutes, walking a long distance (such as 1km), concentrating for 10 minutes, learning a new task like getting to a new place, washing whole body, getting dressed, taking care of household responsibilities, doing day-to-day work, dealing with people they do not know, maintaining a friendship, being emotionally affected by health problems, and joining in community activities. The scale is from 0-4, with 0 being no difficulty, 1 mild, 2 moderate, 3 severe, and 4 cannot do. The scores will be summed to create a cumulative score on a 0-48 scale.

SECONDARY OUTCOMES:
Loneliness/Social Connectedness | Assessed at 0 months after the intervention
  This measure is a standardized index combining five components. First, a 3-item short-form UCLA Loneliness Scale (ULS-3): feeling of lacking companionship, being left out, and isolation (1=Hardly ever, 2=Some of the time, 3=Often; summed). Second, a direct report of loneliness: whether the subject felt lonely last week (1=Yes, 0=No). Third, the Perceived Social Support scale, summing responses to 8 items from Family and Friends subscales (1=Very strongly disagree to 7=Very strongly agree) about emotional support, decision-making help, and sharing joys/sorrows. Fourth, a 2-item Emotional Connection subscale from the Brief Sense of Community Scale, assessing connection to the neighborhood and bond with neighbors (1=Strongly disagree to 7=Strongly agree). Fifth, a single question on the number of close friendships. Measures 1 and 2 are inverted, and all components combined to create an index where higher values indicate greater social connectedness.
Loneliness/Social Connectedness | Assessed at 6 months after the intervention
  The social connectedness measure is a standardized index combining five components. First, a 3-item short-form UCLA Loneliness Scale (ULS-3): feeling of lacking companionship, being left out, and isolation (1=Hardly ever, 2=Some of the time, 3=Often; summed). Second, a direct report of loneliness: whether the subject felt lonely last week (1=Yes, 0=No). Third, the Perceived Social Support scale, summing responses to 8 items from Family and Friends subscales (1=Very strongly disagree to 7=Very strongly agree) about emotional support, decision-making help, and sharing joys/sorrows. Fourth, a 2-item Emotional Connection subscale from the Brief Sense of Community Scale, assessing connection to the neighborhood and bond with neighbors (1=Strongly disagree to 7=Strongly agree). Fifth, a single question on the number of close friendships. Measures 1 and 2 are inverted, and all components combined to create an index where higher values indicate greater social connectedness.
Cognitive function | Assessed at 0 months after the intervention
  Participants will be administered the Mini Mental State Exam. Elders are asked 11 questions and tasks that evaluate various cognitive domains, such as orientation, memory, attention, language, and visuospatial skills. If the question or task is completed correctly, the item receives a score of 1, and 0 otherwise. Scores are summed such that a higher score indicates better cognitive function. The maximum possible score is 30 points.
Cognitive function | Assessed at 6 months after the intervention
  Participants will be administered the Mini Mental State Exam. Elders are asked 11 questions and tasks that evaluate various cognitive domains, such as orientation, memory, attention, language, and visuospatial skills. If the question or task is completed correctly, the item receives a score of 1, and 0 otherwise. Scores are summed such that a higher score indicates better cognitive function. The maximum possible score is 30 points.
Objective Measures of Sleep | Assessed at 0 months after the intervention
  This is a standardized index combining two components comprised of Actigraph device-measured data (subset ~N=1,000): total sleep time and sleep efficiency (asleep time/bedtime). Actigraph data is collected 1 month pre- to 2 months post-intervention. Both measures are combined to form an index, with higher scores indicating better sleep.
Perceived Health Status | Assessed at 0 months after the intervention
  The measure of perceived health status will be a standardized index constructed with two measures. The first measure is self-reported summary of overall health on a scale of 1=Very poor to 5=Very good. The second measures is self-assessed physical pain in the last week on a scale of 0= "no pain" and 10 ="worst pain possible". The second measure of the index will be inverted such that higher values correspond to better perceived health and lower pain.
Perceived Health Status | Assessed at 6 months after the intervention
  The measure of perceived health status will be a standardized index constructed with two measures. The first measure is self-reported summary of overall health on a scale of 1=Very poor to 5=Very good. The second measures is self-assessed physical pain in the last week on a scale of 0= "no pain" and 10 ="worst pain possible". The second measure of the index will be inverted such that higher values correspond to better perceived health and lower pain.
Physical Mobility | Assessed at 0 months after the intervention
  The mobility measure is a standardized index combining three components. First, a self-reported question on whether the elder left home the previous day (1=Yes, 0=No). Second, frequency of engaging in two activities: walking at a moderate pace or floor/stretching/gentle yoga exercises (1=Hardly ever/never to 5=Everyday). Third, a per-day average step count based on Actigraph device data for a subset (~N=1,000). Actigraph measurements are collected from 1 month before to 2 months after the intervention period. When Actigraph data is available, all three measures are combined into an index where higher values indicate greater mobility. If Actigraph data is unavailable, the index is constructed using the first two components.
Physical Mobility | Assessed at 6 months after the intervention
  The measure of mobility will be a standardized index constructed with two measures. The first measure is self-reported mobility question about whether the elder left home the day before, where the responses are either 1 if they did or 0 if they did not. The second measure is a measure of how frequently elders engage in two activities: walking at a moderate pace or floor/stretching/gentle yoga exercises. Responses vary from 1 "Hardly ever/never" to "5 = Everyday". The index is constructed such that an increase in the index corresponds to more mobility.
Agency | Assessed at 0 months after the intervention
  The measure of agency will be measured with a standardized index comprised of two measures. The first measure is a question of the subject's locus of control from the World Values Survey where the subject is asked the extent to which they feel that they have free choice and control over their lives on a scale of 1=No choice at all to 10=A great deal of choice. The second measure is a 2-question subset of the Generalized Self-Efficacy scale that asks about whether the subject feels they can solve most problems with effort and whether they can find several solutions on a scale of 0=No completely to 3=Yes completely. The index is constructed such that an increase in the index corresponds to an increase in agency, capturing higher locus of control and more self-efficacy.
Agency | Assessed at 6 months after the intervention
  The measure of agency will be measured with a standardized index comprised of two measures. The first measure is a question of the subject's locus of control from the World Values Survey where the subject is asked the extent to which they feel that they have free choice and control over their lives on a scale of 1=No choice at all to 10=A great deal of choice. The second measure is a 2-question subset of the Generalized Self-Efficacy scale that asks about whether the subject feels they can solve most problems with effort and whether they can find several solutions on a scale of 0=No completely to 3=Yes completely. The index is constructed such that an increase in the index corresponds to an increase in agency, capturing higher locus of control and more self-efficacy.

OTHER OUTCOMES:
Self-reported Measures of Sleep | Assessed at 0 months after the intervention
  This is a standardized index combining three components. First, self-reported sleep hours based on sleep/wake times. Second, a 7-item Sleep and Insomnia Severity Index assessing the past two weeks: difficulty falling/staying asleep, waking too early (1=None to 5=Very severe), sleep satisfaction (1=Very satisfied to 5=Very dissatisfied), interference with daily function (1=Not at all to 5=Very much), impact on quality of life (1=Not noticeable to 5=Very noticeable), and worry about sleep (1=Not at all to 5=Very much). Third, a Pittsburgh Sleep Quality Index item on overall sleep quality in the past month (1=Very good to 4=Very bad). Measures 2 and 3 are inverted, and all measures are combined to form an index, with higher scores indicating better sleep.
Self-reported Measures of Sleep | Assessed at 6 months after the intervention
  This is a standardized index combining three components. First, self-reported sleep hours based on sleep/wake times. Second, a 7-item Sleep and Insomnia Severity Index assessing the past two weeks: difficulty falling/staying asleep, waking too early (1=None to 5=Very severe), sleep satisfaction (1=Very satisfied to 5=Very dissatisfied), interference with daily function (1=Not at all to 5=Very much), impact on quality of life (1=Not noticeable to 5=Very noticeable), and worry about sleep (1=Not at all to 5=Very much). Third, a Pittsburgh Sleep Quality Index item on overall sleep quality in the past month (1=Very good to 4=Very bad). Measures 2 and 3 are inverted, and all measures are combined to form an index, with higher scores indicating better sleep.
Demand for Intervention Activities | Assessed at 0 months after the intervention
  The demand for interventions measure is an indicator equal to 1 if the subject prefers either intervention (CBT or Group Activities) over a cash transfer in a hypothetical choice, and 0 if they prefer the cash transfer. This comes from a question asking subjects to rank their preference between a Group Activities program, CBT program, or a one-time 1,000 Rs cash transfer.
Demand for Intervention Activities | Assessed at 6 months after the intervention
  The demand for interventions measure is an indicator equal to 1 if the subject prefers either intervention (CBT or Group Activities) over a cash transfer in a hypothetical choice, and 0 if they prefer the cash transfer. This comes from a question asking subjects to rank their preference between a Group Activities program, CBT program, or a one-time 1,000 Rs cash transfer.
Health Management Behavior | Assessed at 0 months after the intervention
  The measure of health management behavior will be comprised of three measures. The first measure is a self-reported question about use of common check-up services in the last 12 months. 1 indicates that the subject did the activity and 0 otherwise. The second measure is a self-report of whether the elder is interested in attending a one-day health camp that is hosted by the research team after the end of the intervention, where subjects can access health measurements such as blood pressure and blood oxygen levels. The third measure is whether the elder actually attended the health camp. The index will be constructed such that an increase in the index indicates more health management behavior.
Health Management Behavior | Assessed at 6 months after the intervention
  The measure of health management behavior will be comprised of one measure. The measure is a self-reported question about use of common check-up services in the last 12 months. 1 indicates that the subject did the activity and 0 otherwise.
Anxiety Score | Assessed at 6 months after the intervention
  Measured using the Generalized Anxiety Disorder 7-item (GAD-7). Scores are constructed by summing answers to 7 questions using a 4-point scale (0=Not at all to 3=Nearly every day, range 0-21). Higher scores indicate more symptoms of anxiety.
Life Satisfaction Score | Assessed at 0 months after the intervention
  Self-reported life satisfaction on a scale (0=Not at all satisfied to 10=Completely satisfied). Note that this measurement taken at 0 months after the intervention is only available for half the sample, collected during the second wave of implementation only.
Life Satisfaction Score | Assessed at 6 months after the intervention
  Self-reported life satisfaction on a scale (0=Not at all satisfied to 10=Completely satisfied). Note that this measurement taken at 0 months after the intervention is only available for half the sample, collected during the second wave of implementation only.
Elder's Caregiver-Elder Relationship Quality Index | Assessed at 0 months after the intervention
  This is a standardized index combining four components. First, we measure of subjective closeness, which is 1 item from the Subjective Closeness Index (SCI) asking "How close do you feel to [caregiver's name]?" with responses ranging from 1=Not at all close to 7=Very close. Second, a measure of relationship strength that is comprised of 4 items from the Relationship Closeness Inventory (RCI) strength subscale, withr responses ranging from 1=Strongly disagree to 7=Strongly agree capturing perceived importance, influence, and mutual understanding in the relationship. Third, we measure communication frequency using one question on how often the caregiver and elder talk about personal concerns, with responses ranging 1=Multiple times a day to 7=Not in the last month). Fourth, we measure perceived burden with 3 items on whether the elder worries about being a burden, hides pain or sickness to avoid worrying the caregiver, or avoids treatment to not burden them, with responses ranging from
Elder's Caregiver-Elder Relationship Quality Index | Assessed at 6 months after the intervention
  This is a standardized index combining four components. First, we measure of subjective closeness, which is 1 item from the Subjective Closeness Index (SCI) asking "How close do you feel to [caregiver's name]?" with responses ranging from 1=Not at all close to 7=Very close. Second, a measure of relationship strength that is comprised of 4 items from the Relationship Closeness Inventory (RCI) strength subscale, withr responses ranging from 1=Strongly disagree to 7=Strongly agree capturing perceived importance, influence, and mutual understanding in the relationship. Third, we measure communication frequency using one question on how often the caregiver and elder talk about personal concerns, with responses ranging 1=Multiple times a day to 7=Not in the last month). Fourth, we measure perceived burden with 3 items on whether the elder worries about being a burden, hides pain or sickness to avoid worrying the caregiver, or avoids treatment to not burden them, with responses ranging from
[Caregiver] Caregiver's Caregiver-Elder Relationship Quality Index | Assessed at 0 months after the intervention
  This is a standardized index composed of three components. First, we measure subjective closeness with 1 item from the Subjective Closeness Index (SCI) asking "How close do you feel to [elder's name]?" with responses ranging from 1=Not at all close to 7=Very close. Second, we measure relationship strength using 4 items from the Relationship Closeness Inventory (RCI) strength subscale, with responses ranging from 1=Strongly disagree to 7=Strongly agree, capturing perceived importance, influence, and mutual understanding in the relationship. Third, we measure communication frequency with 1 item on how often the caregiver and elder talk about personal concerns, with responses ranging from 1=Multiple times a day to 7=Not in the last month. Component 3 is reverse-coded so that higher values indicate a closer and more comfortable relationship between the caregiver and the elder.
[Caregiver] Caregiver's Caregiver-Elder Relationship Quality Index | Assessed at 6 months after the intervention
  This is a standardized index composed of three components. First, we measure subjective closeness with 1 item from the Subjective Closeness Index (SCI) asking "How close do you feel to [elder's name]?" with responses ranging from 1=Not at all close to 7=Very close. Second, we measure relationship strength using 4 items from the Relationship Closeness Inventory (RCI) strength subscale, with responses ranging from 1=Strongly disagree to 7=Strongly agree, capturing perceived importance, influence, and mutual understanding in the relationship. Third, we measure communication frequency with 1 item on how often the caregiver and elder talk about personal concerns, with responses ranging from 1=Multiple times a day to 7=Not in the last month. Component 3 is reverse-coded so that higher values indicate a closer and more comfortable relationship between the caregiver and the elder.
[Caregiver] Caregiver's Well-being Index | Assessed at 6 months after the intervention
  This is a standardized index composed of four components. First, we measure depressive symptoms as the total score on the 9-item Patient Health Questionnaire (PHQ-9), summing responses (0="not at all" to 3="nearly every day", range 0-27). Second, we measure life satisfaction with one question about self-reported satisfaction, with responses ranging from 0=Not at all satisfied to 10=Completely satisfied. Third, we measure caregiving burden, which is the sum of 6 Zarit Burden Scale items on strain and role interference, with responses ranging from 1=Never to 6=Always. Fourth, we measure role and work interference, which is the sum of (1) roles for which caregiving interferes with responsibilities and (2) responses to counterfactual work question ("If you did not have to care for [elder], would you work a lot less, a little less, the same, a little more, or a lot more than you do now?"). The counterfactual is coded 0 = "the same," 1 = "a little less" or "a little more," 2 = "a lot less"
[Caregiver] Caregiver's Well-being Index | Assessed at 0 months after the intervention
  This is a standardized index composed of four components. First, we measure depressive symptoms as the total score on the 9-item Patient Health Questionnaire (PHQ-9), summing responses (0="not at all" to 3="nearly every day", range 0-27). Second, we measure life satisfaction with one question about self-reported satisfaction, with responses ranging from 0=Not at all satisfied to 10=Completely satisfied. Third, we measure caregiving burden, which is the sum of 6 Zarit Burden Scale items on strain and role interference, with responses ranging from 1=Never to 6=Always. Fourth, we measure role and work interference, which is the sum of (1) roles for which caregiving interferes with responsibilities and (2) responses to counterfactual work question ("If you did not have to care for [elder], would you work a lot less, a little less, the same, a little more, or a lot more than you do now?"). The counterfactual is coded 0 = "the same," 1 = "a little less" or "a little more," 2 = "a lot less"
[Meta-Index] Psychological Well-being | Assessed at 0 months after the intervention
  Additionally, to address multiple hypothesis testing, we report effects on three broad outcome domains that group our main outcomes into conceptually related families. The eight primary and secondary outcomes are grouped into three broader domains-psychological well-being, physical health, and cognition. The psychological index is a combination of four indices, described above. (1) Depression score (Geriatric Depression Scale, GDS-15); (2) Functional Impairment Score (WHO-DAS 2.0); (3) Loneliness / Social Connectedness Index; and (4) Agency Index. The first two components will be reverse-coded so that higher values of the index indicate better well-being.
[Meta-Index] Psychological Well-being | Assessed at 6 months after the intervention
  Additionally, to address multiple hypothesis testing, we report effects on three broad outcome domains that group our main outcomes into conceptually related families. The eight primary and secondary outcomes are grouped into three broader domains-psychological well-being, physical health, and cognition. The psychological index is a combination of four indices, described above. (1) Depression score (Geriatric Depression Scale, GDS-15); (2) Functional Impairment Score (WHO-DAS 2.0); (3) Loneliness / Social Connectedness Index; and (4) Agency Index. The first two components will be reverse-coded so that higher values of the index indicate better well-being.
[Meta-Index] Physical Health | Assessed at 0 months after intervention
  To address multiple hypothesis testing, we report effects on three broad outcome domains that group our main outcomes into conceptually related families. The eight primary and secondary outcomes are grouped into three broader domains-psychological well-being, physical health, and cognition. The physical health index is a combination of three indices, described in detail below: (1) Objective measure of sleep (when available); (2) Perceived Health Status; and (3) Physical mobility
[Meta-Index] Physical Health | Assessed at 6 months after intervention
  To address multiple hypothesis testing, we report effects on three broad outcome domains that group our main outcomes into conceptually related families. The eight primary and secondary outcomes are grouped into three broader domains-psychological well-being, physical health, and cognition. The physical health index is a combination of three indices, described in detail below: (1) Objective measure of sleep (when available); (2) Perceived Health Status; and (3) Physical mobility

CONTACTS AND LOCATIONS:
Locations (1):
- JPAL SA at IFMR, Chennai, Tamil Nadu, India